CLINICAL TRIAL: NCT06206993
Title: Effects of Kieser Resistance Training Plus Kieser Pelvic Floor Training vs. Kieser Resistance Training Plus Traditional Pelvic Floor Exercise on Urinary Incontinence in Prostate Cancer Patients After Radical Prostatectomy
Acronym: RECON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Kieser Training Offenbach / Marko Babovic (Unknown); Kieser Training AG Zürich / Dr. David Aguayo (Unknown)
Responsible Party: Principal Investigator, Joachim Wiskemann, Prof. Dr. Joachim Wiskemann, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-458/2019
Record Dates: First submitted 2023-12-15; First posted 2024-01-16 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Prostate Ectomy; Pelvic Floor Disorders; Incontinence, Urinary
Keywords: Prostate Cancer; Pelvic Floor Training; Exercise; Physical Activity; Prostate Ectomy; Incontinence; Cancer; surgery
MeSH Terms: conditions — Prostatic Neoplasms; Pelvic Floor Disorders; Urinary Incontinence; Motor Activity; Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training on the Kieser A5 pelvic floor trainer (Experimental): Participants will receive a supervised full body resistance exercise program with 10-12 machines twice weekly.
  The resistance training for the experimental group includes an intervention program on the Kieser A5 pelvic floor trainer. The training is a predetermined program of the Kieser Training AG. A standardized instruction protocol and custom settings of the seat minimize training or measurement variations. The exercise on the Kieser A5 pelvic floor muscle trainer is standardized and will take 120 s in total which is based on current training theories.
  Interventions: Behavioral: Resistance training including the Kieser A5 pelvic floor trainer
- Resistance training without pelvic floor biofeedback Kieser A5 pelvic floor trainer (Active Comparator): Participants will receive a supervised full body resistance exercise program with 10-12 machines twice weekly.
  Participants in the active comparator group perform the resistance training unit without the pelvic floor biofeedback device A5 and undergo conventional pelvic floor muscle training with a physiotherapist once a week before the resistance training unit starts. Participants are individually informed about the anatomy and function of the pelvic floor muscles and how to correctly contract them. The methodical structure for the movement therapy after prostatectomy suggests that the participants first lay down, then go in the seat, then above the all fours position stand in the upright position tt be treated. Each exercise lasts 3 to 5 min and the session lasts around 20 - 30 min.
  Interventions: Behavioral: Resistance training without pelvic floor biofeedback Kieser A5 pelvic floor trainer

INTERVENTIONS:
Behavioral: Resistance training including the Kieser A5 pelvic floor trainer — In the RECON Study participants of both arms will receive machine-based resistance training. Experimental group will additionally train with Kieser A5 pelvic floor trainer.
  Arms: Resistance training on the Kieser A5 pelvic floor trainer
Behavioral: Resistance training without pelvic floor biofeedback Kieser A5 pelvic floor trainer — In the RECON Study participants of both arms will receive machine-based resistance training. Active Comparator trains without the pelvic floor biofeedback device A5 and undergo conventional pelvic floor muscle training with a physiotherapist once a week before the resistance training unit starts.
  Arms: Resistance training without pelvic floor biofeedback Kieser A5 pelvic floor trainer

SUMMARY:
Surgical removal of the prostate (radical prostatectomy) is the most common therapy in prostate cancer patients. However, urinary incontinence often occurs as a side effect. Although this can recede after a few weeks or months, 12 months after prostatectomy 17 - 34 % of the patients are still incontinent. An effective measure to reduce incontinence is pelvic floor muscle or sphincter training. Various methods exist for this, from pelvic floor gymnastics to training with biofeedback devices and electrical stimulation methods.

Kieser Training, a Germany-wide provider of health-oriented resistance training, has a training device for pelvic floor muscle training. It is a biofeedback device that can be used in public training rooms and does not have to be inserted or glued intimately as with comparable methods. The standardized training program and concept, which allows non-invasive training in public space, has not been evaluated yet.

The aim of the RECON study is to investigate whether Kieser resistance training with integrated Kieser pelvic floor muscle training is as effective as (non-inferior to) Kieser resistance training plus conventional pelvic floor muscle exercise to reduce urinary incontinence in prostate cancer patients after radical prostatectomy. The primary endpoint is the proportion of patients with urinary incontinence at the end of a 12-week training phase (using the 24h pad test). The secondary endpoints are changes in urinary leakage, other incontinence symptoms, incontinence-related quality of life, body composition and changes in strength and overall quality of life.

The design is a two-arm randomized controlled trial with 180 prostate cancer patients. After the initial examination patients will be randomized to one of two groups. Patients in both groups will train for about 60 minutes twice a week for twelve weeks and additionally perform daily tension exercises at home. Patients in group A will perform the resistance training unit with the pelvic floor biofeedback device A5 from the Kieser Training AG and patients of group B will perform the resistance training unit without the pelvic floor biofeedback device A5 and undergo conventional pelvic floor muscle training with a physiotherapist once a week before the resistance training unit starts.

The Recon study will be conducted at the Kieser Training Studio in Offenbach, as a cooperation project of the National Center for Tumor Diseases (NCT), Heidelberg University Hospital and the Kieser Training AG with the Kieser Training franchisee (studio owner) as PhD student at the NCT. The Kieser Training AG is not a sponsor and the study is neither financed nor sponsored.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer
* Radical prostatectomy (inclusion up to three days after discharge from hospital)
* Willingness to train at the exercise facility for 12 weeks, twice per week and to take part in the scheduled testing
* Sufficient German language skills
* Signed informed consent.

Exclusion Criteria:

* Unstable bone metastases or severe cardiac, neurologic, pulmonary or orthopedic diseases which are contraindications to resistance training
* Severe hemorrhoids, anal fissure, or fistulae which are contraindications to pelvic floor muscle training
* Radical perineal prostatectomy (RPP) due to potential pain when using the A5 machine
* Neurological or muscular diseases ruling out successful pelvic floor muscle training
* Pre-surgical incontinence
* Neobladder
* Pacemaker.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 12 of the proportion of continent patients | baseline up to 12 weeks (& 3 month follow-up)
  Major efficacy endpoint (primary endpoint) is the proportion of patients who is continent 12 weeks, with continence defined as no need to wear a pad (1 pads) in the 24 h pad test.
  The International Consultation on Incontinence (organized by the International Consultation on Urological Diseases) recommends that criteria for cure/improve/fail of interventions against urinary incontinence should be based on patient perception as well as objective and semi-objective instruments such as validated questionnaires, diaries and pad tests. In the RECON study, the 24 h pad test will be used as an objective measure of incontinence.

SECONDARY OUTCOMES:
Change from baseline to week 12 in urinary leakage (cumulative pad weight in the 24 h pad test | baseline up to 12 weeks (& 3 month follow-up)
  Cumulative weight of pads with 24h according to the testing procedure below. The International Consultation on Incontinence (organized by the International Consultation on Urological Diseases) recommends that criteria for cure/improve/fail of interventions against urinary incontinence should be based on patient perception as well as objective and semi-objective instruments such as validated questionnaires, diaries and pad tests. In the RECON study, the 24 h pad test will be used as an objective measure of incontinence.
Change from baseline to week 12 in Health related Quality of life, as measured by the EORTC QLQ-C30 | baseline up to 12 weeks (& 3 month follow-up)
  Quality of life will be assessed with the validated 30-item self-assessment questionnaire of the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0). It comprises five multi-item functional scales (physical, role, emotional, cognitive, and social function), three multi-item symptom scales (fatigue, pain, nausea/vomiting), and six single items assessing further symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea) and financial difficulties. Scores range from 0 to 100. A higher score for the functional scales and global health status denote a better level of functioning, whereas a high score for symptom/single-item scale indicate a higher level of symptomatology/problems. Change = (Week 24 Score - Baseline Score)
Change from baseline to week 12 in incontinence related quality of life (EORTC QLQ PSM module) | baseline up to 12 weeks (& 3 month follow-up)
  The prostate cancer module EORTC QLQ PR25 (25-item) is meant for use among patients with prostate cancer varying in disease stage and treatment modality (i.e. surgery, chemotherapy, radiotherapy, etc.) in addition to the QLQ-C30. This instrument contains, among other things, three symptom scales for measuring "bladder symptoms", "intestinal symptoms" and the burden of "incontinence aids". These scales have a value range of 0 to 100 points, with a higher value indicating a higher symptom load.
Change from baseline to week 12 in pain experienced (visual analog scale, VAS) | baseline up to 12 weeks (& 3 month follow-up)
  The visual analogue scale (VAS) entered the realm of pain research in the 1980s, demonstrating a greater sensitivity to increments or decrements in pain than other instruments. It is a subjective pain measurement ranging from "no pain" to "unbearable pain" as two ends of a 10 cm line. The patient marks his subjective sensation on the line. The specified value is then quantified by the investigator. The Reliability of the VAS for acute pain measurement appears to be high
Change from baseline to week 12 in muscle strength (Delfex Sensor System, DSS) | baseline up to 12 weeks (& 3 month follow-up)
  Isometric strength tests will be performed on three resistance training machines by means of a Kieser force sensor. The force sensor is a mobile measuring instrument. During movement, the staking rod of the machine is only moved until the force sensor hits the base plate of the upper weight block from below. By applying additional force, a strain gauge inside the sensor is subjected to elastic bending.
Change from baseline to week 12 in body composition (bioelectrical impedance analysis with the Tanita MC780). | baseline up to 12 weeks (& 3 month follow-up)
  The bioelectrical impedance analyzer Tanita MC780MA will be used for the assessment body composition. A weak electric current is conducted through the body through contacts on hands and feet. Different components of the body act as a resistor (impedance). The measured outcome is the phase angle.

CONTACTS AND LOCATIONS:
Locations (1):
- Kieser Training Offenbach, Offenbach, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No